CLINICAL TRIAL: NCT01480336
Title: The Pharmacokinetics and Electrocardiographic Implications of Adjunctive Amiodarone and Ranolazine Therapy in Patients on Implantable Cardioverter Defibrillators: The Adjunctive Ventricular Arrhythmia Suppression Trial (AVAST) Pilot
Brief Title: The Adjunctive Ventricular Arrhythmia Suppression Trial (AVAST) Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: KLUG003330HE
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Arrhythmia
Keywords: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Amiodarone; Ranolazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amiodarone with Placebo (Placebo Comparator)
  Interventions: Drug: Amiodarone with Placebo
- Amiodarone with Ranolazine (Active Comparator)
  Interventions: Drug: Amiodarone Plus Ranolazine

INTERVENTIONS:
Drug: Amiodarone Plus Ranolazine — Ranolazine 500mg by mouth twice daily
  Arms: Amiodarone with Ranolazine
Drug: Amiodarone with Placebo — stabel dose of amiodarone as prescribed by cardiologist
  Arms: Amiodarone with Placebo

SUMMARY:
The purpose of this study is to learn if combination therapy with amiodarone and ranolazine (an approved drug for chest pain) can help prevent arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ICD who were on a stable dose of amiodarone for the past 60 days

Exclusion Criteria:

* Patients with a life expectancy of less than 6 months
* Patients with moderate or severe hepatic impairment (Child-Pugh Classes B or C) or requiring hemodialysis.
* Pregnancy or lactation.
* Treatment with potent CYP3A inhibitors, including ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, indinavir, and saquinavir
* Treatment with CYP3A inducers, including rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, and St. John's wort.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter Estimates | 12 hours
  Absorption, Peak concentration, time to peak concentration, clearance, area under the curve

SECONDARY OUTCOMES:
Electrocardiogram (ECG) | 12 hours
  The QT/QTc interval and other ECG parameters

CONTACTS AND LOCATIONS:
Overall Officials: William Baker, Pharm.D., Principal Investigator — University of Connecticut
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States